CLINICAL TRIAL: NCT06197997
Title: Strengthening Parenting, Young Children's Social-Behavioral Competence, and Kindergarten Readiness in Schools Serving Low-Income Communities
Brief Title: Resilient, Engaged, and Connected Study
Acronym: REC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00428221; 1R01HD108160-01A1 (NIH)
Record Dates: First submitted 2023-12-07; First posted 2024-01-10 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Parenting; Parenting Intervention
Keywords: Parenting; Chicago Parent Program; CPP

STUDY DESIGN:
Intervention Model Description: The Chicago Parent Program (CPP) is a 12-session group-based parenting intervention designed to strengthen parenting skills and parent engagement in children's learning and improve children's social-emotional and behavioral competence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Title 1 schools receive the Chicago Parent Program intervention (Experimental): The experimental group from Title 1 or Community Schools across two Maryland school districts (Baltimore City Public Schools and Cecil County Public Schools) will receive the Chicago Parent Program intervention.
  Interventions: Behavioral: Chicago Parent Program (CPP)
- Title 1 schools receive the usual school practice (No Intervention): The control group from Title 1 or Community Schools across two Maryland school districts (Baltimore City Public Schools and Cecil County Public Schools) will receive the usual school practice.

INTERVENTIONS:
Behavioral: Chicago Parent Program (CPP) — The Chicago Parent Program (CPP) is a 12-session group-based parenting intervention designed to strengthen parenting skills and parent engagement in children's learning and improve children's social-emotional and behavioral competence.
  Arms: Title 1 schools receive the Chicago Parent Program intervention

SUMMARY:
Purpose of this study is to test the effectiveness and implementation of an evidence-based parenting intervention for improving parenting and school outcomes in a sample of 4-year-old children enrolled in public prekindergarten (PreK) programs in Maryland.

DETAILED DESCRIPTION:
Using a hybrid Type 2 effectiveness-implementation design, this study tests the effectiveness and implementation of an evidence-based parenting intervention for improving parenting and school outcomes in a sample of 4-year-old children enrolled in public prekindergarten (PreK) programs in Maryland. Thirty Title 1 schools across two Maryland school districts (Baltimore City Public Schools n=20; Cecil County Public Schools n=10) will be randomized into experimental (receive the Chicago Parent Program intervention) or control (usual school practice) conditions. The Chicago Parent Program (CPP) is a 12-session group-based parenting intervention designed to strengthen parenting skills and parent engagement in children's learning and improve children's social-emotional and behavioral competence. All schools will participate for 2 years. In the experimental condition, school staff trained in CPP will implement the program in groups of 10-15 parents of PreK students in a virtual group or in-person group format (format order counterbalanced). Parents in the control condition will complete surveys only. Study outcomes for all participants will be evaluated at PreK baseline (T1), 4-5 months post baseline (T2), in the fall of kindergarten (T3), and at the end of kindergarten (T4). Outcomes include children's social-emotional-behavioral competence, parent engagement in early childhood education, and parenting skills; school community cohesion; kindergarten readiness, chronic absence, and retained in kindergarten. Additional evaluation data will be collected in the experimental condition assessing perceived effectiveness, implementation quality, uptake, and cost-effectiveness to understand factors that affect the likelihood the program can be successfully integrated and sustained in urban and rural school settings. Demographic background variables will be collected from parents at baseline. Variables include the caregiver role in relation to the PreK child; the race, ethnicity, age, and gender of the parent and PreK child; primary language spoken in the home; and parents' education, employment status, marital status, and annual household income. The investigators will also assess nine family economic hardships experienced over the past 12 months. Demographic background variables will also be collected from PreK teachers at baseline and K teachers in the fall of K and will include gender, age, race, ethnicity, education, and teaching experience at the teacher's current school.

ELIGIBILITY:
Inclusion Criteria:

Title 1 public school or Community School in Cecil County or Baltimore City, or located in a community designated as high need by the Maryland State Department of Education based on a score of 0.6 on the Center for Disease Control Social Vulnerability Index:

* has at least 1 full-day public PreK classroom with 20+ students;
* school has not previously offered CPP;
* principal consents to being randomized and participate for 2 years;
* principal consents to study team recruiting parents, teachers, and staff to participate in the study.

PreK Parents:

* Parent (biological, step, adoptive, foster), grandparent, or legal guardian of 4-5 year old student enrolled in participating PreK program;
* 18+ yrs;
* speaks English or Spanish;
* consents to allowing access child's school identification.

Teachers:

* PreK or K teacher in classroom of student of participating parent;
* consents to completing study surveys.

CPP Group Leaders:

* completes CPP group leader training
* agrees to lead CPP groups
* speaks English or Spanish
* at least a High School diploma/General Equivalency Diploma (GED)
* consents to completing surveys and submitting audio recorded CPP sessions for fidelity assessment

School-based personnel inclusion criteria:

* Principal, teacher, or other school-based staff involved in CPP implementation
* consents to interview on perspectives about CPP in the school

Exclusion Criteria:

* Principal cannot commit staff to offering CPP groups
* school previously offered CPP
* school located in a geographic area with less than 80% connectivity
* PreK Parents previously participated in CPP
* Teachers: teacher also a participating parent or CPP group leader
* School-based personnel: Principal, teacher, or other school-based staff is a study parent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Social-behavioral readiness as assessed by the social-behavioral domain of the Kindergarten Readiness Assessment (KRA). | 1-year follow-up
  School district's measure of children's social-behavioral readiness to learn at kindergarten entry. Kindergarten Readiness Assessment (KRA) assesses 4 domains of readiness. Domain scores range from 202-298. Higher score is a better outcome.
Percentage of children who reported chronic absence | 1 year
  Percent of children missing 10% or more school days during the kindergarten year. Data will be collected on number of days the school district records the students as absent from school.
Percentage of children who retained in grade | 1 year
  Percentage of children retained in kindergarten for another year. Data will be collected based on report from the school district on whether child was retained.
Social Competence and Behavior Evaluation (SCBE-30) score (Teacher Version) | Baseline, post-intervention up to 4 months, post-intervention up to 8 months, 1-year follow-up
  change in measures of children's behavior and social-emotional skills from perspective of teachers. Teachers complete the Social Competence and Behavior Evaluation (SCBE-30). Teacher version contains 3 sub scales of 10 items each. Subscale scores range from 10- 60. Higher scores indicate higher levels of social competence.
Social Competence and Behavior Evaluation (SCBE-30) score (Parent Version) | Baseline, post-intervention up to 4 months, post-intervention up to 8 months, 1-year follow-up
  change in measures of children's behavior and social-emotional skills from perspective of parents. Parent version of the SCBE-30 contains 3 sub scales of 10 items each. Subscale scores range from 10- 60. Higher scores indicate higher levels of social competence.
Eyberg Child Behavior Inventory (ECBI) score | Baseline, post-intervention up to 4 months, post-intervention up to 8 months, 1-year follow-up
  change in child behavior problems on the Eyberg Child Behavior Inventory (ECBI) ECBI contains two sub scales of 36 items each; Intensity Scale scores can range from 36-252; Problem Scale scores can range from 0-36. Higher scores indicate worse outcomes.
Parent engagement as assessed by the Parent-Teacher Involvement Questionnaire | Baseline, post-intervention up to 4 months, post-intervention up to 8 months, 1-year follow-up
  change in measures of parent's engagement in their children's early education from the perspective of teachers. Teachers will compete a 7-item measure of parent engagement from the Parent-Teacher Involvement Questionnaire. Scores range from 7-35. Higher scores indicate more parental involvement.
Parent engagement as assessed by the Parent Engagement in Early Childhood Education (PEECE) Survey | Baseline, post-intervention up to 4 months, post-intervention up to 8 months, 1-year follow-up
  change in measure of parent engagement on the Parent Engagement in Early Childhood Education (PEECE) Survey, a 25-item measure of parent engagement. Scores can range from 25-100. Higher scores indicate higher involvement.

SECONDARY OUTCOMES:
Total kindergarten readiness score | 1 year
  Total kindergarten readiness score as assessed by the Kindergarten Readiness Assessment including language/literacy, numeracy skills, physical well-being/motor development, and social-behavioral readiness. Administered by and calculated by the school district.
Parenting skills as assessed by the Parenting Questionnaire | Baseline, post-intervention up to 3 months, 1-year follow-up
  change in parenting skills measured by the Parenting Questionnaire a measure of parents' use of positive discipline, harsh discipline, and consistency of discipline techniques. The score ranges from 40-200. There are 3 subscales of interest for the parenting questionnaire that include: (1) Warmth: higher scores = greater warmth; (2) Corporal Punishment: higher scores = greater use of corporal punishment, and (3) Following Through on Discipline: higher scores = more likely to follow through on discipline.
Social connectedness as assessed by Intervention Group Environment Scale | post-intervention up to 4 months
  Measures parents' sense of belonging and connection with the school, using the 25-item Intervention Group Environment Scale and items are measured along a 5-point continuum of strongly disagree to strongly agree. Includes 3 sub scales. Scores can range from 0-5 with higher scores indicating greater social connectedness.
Parent Satisfaction as assessed by the Chicago Parent Program Satisfaction form | Post-intervention up to 4 months
  Measured using the Chicago Parent Program Parent Satisfaction Form. The survey Includes 16 items. Scored on a Likert-type scale, aspects of the program that were most and least beneficial, and the extent to which the participant would recommend the program to other parents. Each item is scored and interpreted separately.
CPP Reach as assessed by percent of eligible parents enrolled | At baseline
  CPP Reach is defined by parent participation in CPP and will be measured by percent of eligible parents enrolled.
CPP Effectiveness as assessed by End of Program Satisfaction score | Immediately post intervention
  Parents will complete the End of Program Satisfaction Form at post-intervention to assess their satisfaction of the extent to which CPP improved their parenting skills, their children's behavior, their confidence in supporting their children's school success; supported their relationships with their children's teacher and school; created challenges for participation (including technology challenges for virtual groups and transportation challenges for in person groups); and their overall satisfaction with CPP. 8 questions on a 4-point scale, 8 questions on a 3 point scale, and 4 open questions. Each item analyzed separately, higher scores indicate higher satisfaction.
CPP Perceived effectiveness as assessed by qualitative interview | Immediately post-intervention (intervention group)
  Perceived effectiveness will also be assessed from interviews with principals, school staff, and CPP group leaders (approximately 4 total individuals from each school) to understand their perceptions of CPP's benefits and limitations.
CPP Adoption as assessed by qualitative interview | Immediately post-intervention (intervention group)
  CPP Adoption will be assessed from interviews with school staff involved in CPP implementation (i.e., CPP group leaders, school leadership - approximately 4 total individuals from each school) to understand whether and how CPP was folded into their normal workflow; perceived benefits and challenges with offering virtual versus in-person CPP; what the participant learned over the course of the two years of implementation; whether the participant would want to adopt CPP at their school and why; and if CPP were to continue at their school, what the participant believes is needed to make CPP work well for the participant.
Percentage of CPP group-leader retention rate | 2 years
  The investigators will collect data on group leader retention over two years
CPP Implementation challenges as assessed by qualitative interview | 2 years
  Differences in implementation challenges by rural versus urban school districts (e.g. travel distance to school, space in schools) and virtual versus in person groups (e.g. ease of internet access, space in schools).
Social Connectedness in Group Environments Scale (Parent) | Immediately post-intervention (intervention group)
  Parent data will include CPP parent ratings of social connectedness formed within their group as measured by the Social Connectedness in Group Environments Scale. This is a 25-item parent report survey with 3 subscales measuring parents' perceptions of cohesion and sense of belonging among group members, extent to which group leaders generated a positive group environment and negative interactions among group members. Items are scored on a 5-point scale of strongly agree to strongly disagree. Score range 25-125. Higher score greater social connectedness.
Percentage of parents who completed CPP | Immediately post-intervention (intervention group)
  CPP dose (number of sessions attended and CPP practice assignments completed) will be collected based on the session reports.
Quality of Parents' Participation in the CPP groups as assessed by the Quality of Participation score | Immediately post-intervention (intervention group)
  This will be assessed after the 11th session by group leaders using the Quality of Participation Form (QPF). The QPF is a 7-item group-leader report of the extent to which parents are actively engaged in the group sessions supportive to other members in the group, open to trying to new strategies, and able to correctly apply program principles, and quality of parent participation in the CPP groups. Items are rated from 1 (not at all) to 4 (most of the time) and summed. Score range 7-28, higher score better quality.
CPP Implementation Quality as assessed by CPP Fidelity Checklist score | Up to 12 weeks
  This will be assessed by independent raters from a random selection of three audio-recorded CPP sessions per 12-session group using the CPP Fidelity Checklist developed by the study team members. The CPP Fidelity Checklist assesses group leader competence (skill) and adherence to the protocol. For competence, there are 16 items (score range 1-3). For adherence, there are 12-14 items scored yes/no, and the score ranges from 0 to 100 percent adherence. Higher scores indicates better fidelity adherence.
Maintenance of CPP as assessed by implementation costs | Immediately post-intervention (intervention group)
  Maintenance is defined as the likelihood of schools being able to sustain CPP. Data will include CPP implementation costs of in-person versus virtual CPP groups (including the Conditional Cash Transfers for participating in the CPP groups).
Maintenance of CPP as assessed by qualitative interview | Immediately post-intervention (intervention group)
  Maintenance is defined as the perceived likelihood of schools being able to sustain CPP based on the interviews with school-based staff (approximately 4 total individuals from each school).

OTHER OUTCOMES:
Cost-effectiveness | Post-intervention up to 3 months
  Cost of the intervention will be estimated using incremental cost effectiveness ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Gross, DNSc, Principal Investigator — JHU School Of Nursing
Locations (2):
- United States (2):
  - Johns Hopkins School of Nursing, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Parent and teacher de-identified survey data will be available for limited data sharing. Interview and fidelity data will not be shared due to difficulties fully de-identifying the transcripts. Student administrative data will not be shared due to data sharing restrictions associated with the Family Educational Rights and Privacy Act.
Supporting Information: Study Protocol
Time Frame: At the conclusion of the study

REFERENCES:
- [Derived] Gross D, Breitenstein SM, Jeon L, Perrin N, Shen K, Bettencourt AF. Resilient, engaged and connected (REC) study: protocol for a type 2 cluster-randomised trial of the Chicago Parent Program in prekindergarten in low-income urban and rural communities. BMJ Open. 2025 Apr 17;15(4):e099204. doi: 10.1136/bmjopen-2025-099204. PMID 40246571